CLINICAL TRIAL: NCT01116310
Title: Randomized, Double-blind, Placebo-controlled Clinical Trial, to Evaluate the Efficacy and Tolerability of the Combination of Soy Isoflavones and Red Clover Extract (FITOGYN) in the Treatment of the Hot Flushes in Menopausal Women.
Brief Title: Clinical Trial to Evaluate the Efficacy of FITOGYN Versus Placebo on the Vasomotor Symptomatology Associated With Menopause
Acronym: TRYSEM
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Laboratorios Casen-Fleet S.L.U. (Industry)
Collaborators: Apices Soluciones S.L. (Industry); Asociacion Colaboracion Cochrane Iberoamericana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LCF-GIN-2008-EC02
Record Dates: First submitted 2010-05-03; First posted 2010-05-04 (Estimated); Last update posted 2011-09-28 (Estimated); Status verified 2011-09

CONDITIONS: Postmenopausal Women With Moderate Vasomotor Symptoms
Keywords: Hot flushes; Hot flashes; menopause; postmenopause; Soy isoflavones; Red clover; Equol
MeSH Terms: conditions — Hot Flashes | interventions — Soybean Proteins

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fitogyn (Experimental): 4 weeks with placebo followed by 16 weeks with Fitogyn, both taking two capsules per day during the breakfast.
  Interventions: Drug: Soy isoflavones (Glycine max L) and red clover extract (Trifolium pretense L); Drug: Placebo
- Placebo (Placebo Comparator): 20 weeks with placebo, taking two capsules per day during the breakfast.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Soy isoflavones (Glycine max L) and red clover extract (Trifolium pretense L) — Bottles containing 60 capsules, 53.5 mg/capsule of isoflavones
  Other Names: Fitogyn
  Arms: Fitogyn
Drug: Placebo — Bottles containing 60 capsules.

SUMMARY:
The purpose of this study is to evaluate the efficacy of FITOGYN vs. placebo on the vasomotor symptomatology associated with menopause, to evaluate the symptoms of anxiety, the metabolic parameters in menopause and to evaluate the quality of life associated to the vasomotor symptoms of menopause.

DETAILED DESCRIPTION:
One of the most significant problems for assessing treatment of hot flushes is the placebo effect. A Phase IV study with an innovative design, intended to additionally assess such effect, is reported. The efficacy of Fitogyn for the treatment of hot flushes in menopausal women with moderate symptoms will be assessed. Secondary objectives will include evaluation of the impact of Fitogyn as compared to placebo on overall menopause symptoms (fatigue, joint pain, vaginal dryness, and sleep disturbances), anxiety, quality of life, and cardiovascular parameters. Equol levels in blood will also be measured to study its potential impact on the outcome of treatment with these isoflavones.

The duration of the study participants will be 22 weeks. 7 visits are planned during the study:

After the screening visit (visit 1), women selected will report on the daily occurrence of hot flushes for 2 weeks without treatment. If they experience the required number of hot flushes (35-70 hot flushes in the prior week and 9 or more of them with at least moderate intensity), a 4-week placebo run-in period will start (visit 2). After this time (Visit 3), women with a decrease lower than 25% in the number of hot flushes and a treatment adherence of at least 80% will be randomised to receive treatment (Fitogyn vs placebo) for 16 weeks.

During visit 3, baseline assessments of primary and secondary variables will be carried out. Additionally, blood and urine samples will be obtained to conduct hematological and biochemical tests, and assess thyroid function and lipid profile. In addition, patients will complete the following scales: "Menopausal Rating Scale (MRS)", the scales of anxiety (HADS) and quality of life (Scale of Cervantes).

Visits 4, 5 and 6: To assess every 4 weeks the treatment adherence, to do a safety evaluation and daily collection of hot flashes.

Visit 7: End of study (week 22 of study). During this visit the same activities described for visit 3 will be performed.

SUBSTUDY:

TITLE: "Evaluating the impact of the combination of soy isoflavones and red clover extract (FITOGYN) compared to placebo on some markers of atherogenesis"

The substudy will be conducted in a subsample of approximately 90 patients and will involve those Investigational Sites willing to conduct the substudy, given that they have the means for the proper and correct handling of samples. This study has an exploratory purpose, and will provide useful insight into the specific mechanisms of action of phytoestrogens as well as generate new hypotheses that can guide future research on this product. Additionally, blood equol levels will be measured to study their potential effect on treatment outcome with these isoflavones.

A number of biological parameters have been identified that are clearly related to the process of atherogenesis. This measurement would be from blood collections performed at baseline and the end of the trial, so that new blood collections will not be necessary beyond those already planned.

The selected parameters are:

1. Level of insulin resistance from HOMA.
2. Low density lipoprotein (LDL), oxidized (ox LDL) concentration.
3. Asymmetric dimethyl arginine concentration in endothelial cell culture
4. Measure the ratio of prostacyclin / thromboxane in urine.
5. Genesis of tissue factor in the endothelium.
6. Measurement of blood levels of equol.

ELIGIBILITY:
Inclusion Criteria:

* Women between 45 and 60 years of age.
* Women in, the immediate or established postmenopausal phase, defined as women with: a) 12 months or more spontaneous amenorrhea or b) 6 months or more spontaneous amenorrhea with levels of follicular stimulating hormone (FSH) above 40 mIU / ml.
* Women with between 35 and 70 episodes of hot flashes (9 or more hot flashes should be of at least moderate intensity) in the week prior to the pre-inclusion period with placebo
* Women who have given written informed consent.

Exclusion Criteria:

* Women with surgical menopause.
* Treatment with HRT within 6 months of the screening visit.
* Patients who needs oncological or immunosuppressive treatment during the expected follow-up period.
* Patient with difficult follow-up or with psycho-neurological problems that hinder proper assessment (alcoholism, depression not caused by menopause, etc.)
* Patients who, at the discretion of the investigator, can not be evaluated according to criteria established in this protocol
* Patients following a vegetarian diet
* Patients with any relevant gastrointestinal disease
* Patients with a prior diagnosis of hypothyroidism or other clinically relevant thyroid disorder.
* Patients treated and / or diagnosed or with suspicion of cancer.
* Patients with diabetes mellitus who require insulin therapy.
* Patients with current diagnosis of an affective disorder (e.g. depression), anxiety disorder, or psychotic disorder.
* Patients with an organic mental disorder
* Patients with neuropathic pain or any other form of pain that receive or need treatment with antidepressives or anticonvulsivants.
* Patients receiving or requiring treatment with antidepressives or anticonvulsivants for other motives (for example, prevention of the migraine).
* Patients consuming more than 2 alcoholic drinks (16-20 gr.) per day
* Patients who have been treated with antibiotics within 3 months of the screening visit.
* Patients receiving or requiring treatment with clonidine or vitamin E.
* Patients who are treated with NSAIDs
* Patients allergic to any of the components of FITOGYN
* Patients who took less than 80% of the capsules in the pre-inclusion period with placebo.
* Patients whose weekly number of hot flushes is reduced by 25% or more during the pre-inclusion period as compared to the week prior to the initiation of that period.

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 166 (Estimated)
Dates: Start 2010-04; Primary Completion 2012-05 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Mean Change in the number of symptoms of hot flashes (including night sweats) at the end of the study (week 22) with respect to baseline (week 6). | 16 weeks
  This change will be expressed in absolute value and proportion of reduction with regard to the number basal of symptoms reported in the last week of the period of pre inclusion. The average or average of the reduction of hot flushes in every week of treatment and at the end of the treatment will be compared. This information will be obtained for every group and recorded by the women using a "hot flushes diary".
  Additionally, the average change will be evaluated using the hot flash score (frequency combined with intensity) following the same methodology.

SECONDARY OUTCOMES:
Intensity of Hot Flashes | 16 weeks
  Intensity of the hot flushes that the participants communicate in the "hot flushes diary". The variable "intensity" of symptoms will be gathered in the categories of "mild", "moderate", "intense" and "very intense ", according to Sloan et al. J clin Oncol. 2001 dec 1;19 (23):4280-90 definitions.
Impact of the treatment with FITOGYN on the overall symptoms of menopause: fatigue, joint pain, vaginal dryness and sleep disturbances among others. | 16 weeks
  The information about symptoms of the menopause will be gathered across Heinemann's Menopause Rating Scale (Self-administered instrument that evaluates 11 symptoms of menopause on a 5-point scale from 0, no symptom, to 4, extremely severe symptom. The total score includes 3 dimensions or factors: psychological, somato-vegetative, and urogenital. The overall score will be obtained for each domain and assessed at baseline and after 16 weeks of treatment.)
Effect of the treatment with FITOGYN in the level of anxiety of postmenopausal women. | 16 weeks
  The anxiety subscale of the Hospital Anxiety-Depression Scale (HADS) will be used. HADS is a self-administered instrument comprised of 14 items (7 explore symptoms of depression and 7 others explore symptoms of anxiety). Each item is scored from 0 to 3 where 0 represents no symptom and 3 the most severe or frequent symptoms. Two scores are obtained by summing the 7 items of each sub-scale, depression and anxiety (HADS-D and HADS-A), with a score range for each from 0 to 21. The overall score will be obtained and for the anxiety domain assessed at baseline and after 16 weeks of treatment.
Effect of the treatment with FITOGYN in the quality of life of postmenopausal women. | 16 weeks
  The Scale of Cervantes will be used to evaluate quality of life. It consists of 31 items that are distributed in the following dimensions:
  * Menopause and health (15 items assessing vasomotor symptoms, health and aging)
  * Sexuality (4 items)
  * Relationships (3 items)
  * Psychic domain (9 items) The overall score will be obtained and assessed for each domain at baseline and after 16 weeks of treatment.
Evaluate the change in the subject's lipidic profile. | 16 weeks
  The average difference in mm/dL between baseline and after 16 weeks of treatment will be determined.
Evaluation of the safety and tolerability. | 16 weeks
  The average difference between baseline and after 16 weeks of treatment in some haematological (Haemoglobin, WBC Differential Count and platelets), biochemistry (standard biochemistry witch include at least Lactate dehydrogenase, cholesterol, triglycerides and thyroid function) and urinalysis parameters will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Joaquím Calaf, Dr., Study Chair — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau; Cano Antonio, Dr., Study Chair — Hospital Doctor Pesset
Locations (20):
- Spain (20):
  - Hospital Central de Asturias, Asturias
  - Hospital del Cruces, Barakaldo
  - Assir CAP Sant Martí, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - USP Instituto Universitario Dexeus, Barcelona
  - ASSIR CAP San Andreu, Barcelona
  - Hospital Universitari Vall d'Hebrón, Barcelona
  - Hospital Monteprincipe, Boadilla Del Monte, Madrid
  - Hospital General de Ciudad Real, Ciudad Real
  - Centro Diatros, Gavá (Barcelona)
  - Hospital Universitario de Guadalajara, Guadalajara
  - Consorci Sanitari d l´Anoia-H. de Igualada, Igualada, Barcelona
  - Centro de Estudios de Obstetricia y Ginecología Asociado Lugo, Lugo
  - Gabinete Médico Velázquez, Madrid
  - Instituto Palacios, Madrid
  - Hospital Mateu Orfila, Maó
  - H. San Joan d'Alacant, San Juan, Alicante
  - Hospital Universitario La Fe, Valencia
  - Hospital Doctor Pesset, Valencia
  - Hospital Miguel Servet, Zaragoza